CLINICAL TRIAL: NCT07297953
Title: Access Sheath and stENT Trial
Acronym: ACCENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Khurshid Ghani, Clinical Professor of Urology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00264257
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stone; Ureteral Stone
Keywords: Ureteral stent; Ureteroscopy and lithotripsy; Surveys; Quality of life
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be informed of the presence or absence of a stent immediately following participants surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stent omission arm (Other): Participants will complete surveys before and after a planned ureteroscopy and lithotripsy for stone disease.
  Interventions: Other: Surveys
- Stent placement arm (Other): Participants will complete surveys before and after a planned ureteroscopy and lithotripsy for stone disease.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — Surveys will be completed for each group at the following timeframes: baseline (pre-procedure, daily up to 7-10 days or until stent is removed (if placed), 30 days after the procedure. Additionally, participants medical records will reviewed for information.

SUMMARY:
The study is being completed to compare patient reported outcomes for stent omission vs. placement after using a ureteral access sheath for uncomplicated ureteroscopy.

Participants that consent for the study will complete baseline PRO questionnaires. A UAS will be used during surgery, and the size left to the discretion of the surgeon. At the end of the procedure, the urologist will evaluate the ureter for iatrogenic injury, and the ureter will be graded using the Post Ureteroscopic Lesion Scale (PULS). Patients assessed with PULS 0 and PULS 1 will meet 2nd stage eligibility and will be randomized 1:1 to either stent omission or stent placement. When a stent is placed, the stent type and decision to leave a string (tether) will be at the operating urologist's discretion.

Hypothesis:

- stent omission arm will be non-inferior to stent placement in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference and Pain Intensity, and have lower 30-day healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Planned ureteroscopy using a Ureteral Access Sheath (UAS) for treatment of unilateral kidney and/or ureteral stones in patients that have an existing ureteral stent (pre-stented)
* Planned treatment of unilateral renal and/or ureteral stones, in a single procedure.
* Renal stone defined as only renal location of stone(s)
* Ureteral stone defined as ureteral only location of stone(s)
* Ureteral and renal stone(s)
* No evidence of significant ureteral injury on intra-operative assessment (Post-Ureteroscopy Lesion Scale (PULS) Grade 0 or 1)
* Ability and willingness to complete and adhere to survey questions and responses throughout study duration.

Exclusion Criteria:

* Pregnancy
* Ureteric injury during ureteroscopy (PULS ≥ Grade 2)
* Evidence of ureteral stricture
* Anatomical abnormalities (e.g., solitary, horseshoe, fused crossed ectopia, pelvic kidney, urinary diversion)
* Known planned secondary or staged procedure
* Indwelling nephrostomy tube
* Bilateral ureteroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Differences in PROMIS Pain Interference | Baseline (before procedure), 7-10 days after procedure
  This is a 6-item survey which participants select a response for each item from 1=not at all to 5=very much for how much pain interfered with their life. The scores range from 6-30 with a higher score indicating greater interference.

SECONDARY OUTCOMES:
Differences in PROMIS Pain intensity | 7-10 days after procedure
  This is a 3-item survey which participants select a response for each item from 1=no pain to 5=very severe for intensity of their pain. The scores range from 3-15 with a higher score indicating greater pain intensity.
Differences in PROMIS Pain intensity | 4-6 weeks after procedure
  This is a 3-item survey which participants select a response for each item from 1=no pain to 5=very severe for intensity of their pain. The scores range from 3-15 with a higher score indicating greater pain intensity.
Differences in Urinary Symptoms based on the Lower Urinary Tract Dysfunction Research Network (LURN) Symptom index (SI)-10 | 7-10 days after procedure
  The LURN SI-10 (10-Item LURN Symptom Index) assesses urinary frequency, nocturia, urgency, incontinence, bladder pain, voiding and post-micturition symptoms. Responses for each item range from 0 to 4 or 0 to 3 and are then summed for total scores ranging from 0 to 38 (higher scores = worse symptoms/bother).
Differences in Urinary Symptoms based on the Lower Urinary Tract Dysfunction Research Network (LURN) Symptom index (SI)-10 | 4-6 weeks after procedure
  The LURN SI-10 (10-Item LURN Symptom Index) assesses urinary frequency, nocturia, urgency, incontinence, bladder pain, voiding and post-micturition symptoms. Responses for each item range from 0 to 4 or 0 to 3 and are then summed for total scores ranging from 0 to 38 (higher scores = worse symptoms/bother).
Difference in PROMIS Social Roles & Activities | Daily after procedure (10 days or up to stent removal)
  This is one question from the PROMIS that participants select from Never (5) to Always (1) whether there is trouble doing all of participant's usual work. A lower score indicates more trouble.
Difference in Pain intensity assessment based on the Visual analog scale | Daily after procedure (10 days or up to stent removal)
  Participants pain level is selected from 0-10 with a higher score indicating greater pain.
Treatment Satisfaction based on the International Consultation on Incontinence Questionnaire Short Form (ICIQ-S) | 7-10 days post procedure and 4 weeks
  This is a 6-item questionnaire that participants complete regarding the satisfaction with treatment. The range of scores for each question is between 0-5, with a range of score between 0-24 with a higher score indicating greater satisfaction.
Count of days off work Patient | Day 7 post procedure and 4 weeks post procedure
Count of days off work Caregiver | Day 7 post procedure and 4 weeks post procedure
Composite healthcare utilization metric within 30 days (WinRatio) | Up to 30 days after procedure
  WinRatio composite healthcare utilization score ranges from 1 to 6 based on each participants highest level of healthcare utilization, with higher score indicating a worse outcome: 6) Hospitalization and ICU care; 5) Unplanned hospitalization; 4) Additional OR or Interventional Radiology procedure 3) Emergency department visit; 2) Ambulatory encounter: clinic visit or diagnostic outpatient testing; 1) Ambulatory encounter: phone call or electronic medical record.
Abnormal imaging findings within 60 days | within 60 days of procedure
  Urological imaging performed within 60 days per surgeon or patient preference.
Stone-free rates within 60 days | within 60 days of procedure
  X-ray, Ultrasound, computerized tomography (CT) scan, or any combination
Differences in PROMIS Pain Interference | 4-6 weeks after procedure
  This is a 6-item survey which participants select a response for each item from 1=not at all to 5=very much for how much pain interfered with their life. The scores range from 6-30 with a higher score indicating greater interference.

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid Ghani, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No